CLINICAL TRIAL: NCT00665483
Title: Design of Optimally-diagnostic Skin Test Solutions for Diagnosis of Sensitisation to a 6-grass Pollen Mixture, House Dust Mite (Dermatophagoides Pteronyssinus), Birch Pollen, and Mugwort Pollen
Brief Title: Design of Optimally-diagnostic Skin Test Solutions for Diagnosis of Sensitisation to a Pollen and Dust Mite Mixture.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: AL0205PR; 2006-005304-14 (EudraCT Number)
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Type I Allergy
MeSH Terms: interventions — Patch Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Skin Prick Test
  Interventions: Other: Skin Prick Test

INTERVENTIONS:
Other: Skin Prick Test — Skin Prick Test

SUMMARY:
Multicenter Skin Prick Test

ELIGIBILITY:
Inclusion Criteria:

* anamnesis referring to suspicion of an IgE-mediated allergy
* positive Skin Prick Test in the medical history to at least one of the investigational allergens with an existing anamnesis

Exclusion Criteria:

* serious chronic diseases
* Other perennial allergies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2007-03; Primary Completion 2007-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Optimal trade-off between sensitivity and specificity | December 2007 - December 2008

SECONDARY OUTCOMES:
Evaluation of the documentation of adverse events | January - December 2008

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Wagner, MD, Principal Investigator — Klinikum Darmstadt
Locations (1):
- Klinikum Darmstadt, Darmstadt, Hesse, Germany

REFERENCES:
- See also: Leader in specific allergy research and therapy — http://www.allergopharma.de
- See also: Click here for information about this trial in the European Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/trial/2006-005304-14/DE